CLINICAL TRIAL: NCT03178461
Title: The Effect of Warmed Parenteral Fluids During Vaginal Delivery and Cesarean Section
Brief Title: The Effect of Warmed Parenteral Fluids During Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, hanoch schreiber, Dr, Meir Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0049-17-MMC
Record Dates: First submitted 2017-05-30; First posted 2017-06-07 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Delivery, Obstetric
Keywords: Caesarean Section; Delivery

STUDY DESIGN:
Intervention Model Description: Randomization two 2 groups according to temperature of IV fluids. One group will receive room temperature fluids and the other group will receive body temperature fluids.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Room temperature parenteral fluids (No Intervention): This group will receive IV room temperature fluids, which is the standard of care.
  The composition of the fluids given will be normal saline with 5% dextrose.
- Body temperature parenteral fluids (Experimental): This group will receive IV warmed fluids, body temperature, which is the experimental intervention.
  The composition of the fluids given will be normal saline with 5% dextrose.
  Interventions: Other: Body temperature parenteral fluids

INTERVENTIONS:
Other: Body temperature parenteral fluids — 2 study groups shall receive the same parenteral fluids but at different temperatures.
  Arms: Body temperature parenteral fluids

SUMMARY:
To evaluate the influence of warm IV fluids during delivery and cesarean section on perinatal outcomes.

DETAILED DESCRIPTION:
Prospective randomized controlled trial. Assessing the influence of warmed parenteral fluids during delivery/cesarean section on the obstetrical and neonatal outcome. The investigators will randomize parturients during the active phase of labor to receive either body temperature warmed parenteral fluids or room temperature parenteral fluids. Both groups will receive the same fluid composition of 5% dextrose with normal saline. The investigators will compare the obstetrical and neonatal outcomes of the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies
* term pregnancies
* receiving parenteral fluids

Exclusion Criteria:

* high order pregnancies
* preterm pregnancies (before 37 weeks of gestation)
* known fetal major anomaly
* known fetal significant chromosomal/genetic abnormality

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only females are pregnant. The baby can be of either sex
Enrollment: 7000 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Length of the second stage of labor | up to 5 hours from complete cervical dilation
  How much time did it take from complete cervical dilation to the delivery of the baby.

SECONDARY OUTCOMES:
Prevalence of perineal tears and episiotomies | immediately after vaginal birth
  The prevalence of perineal tears and episiotomies that occurred during vaginal delivery
Neonatal APGAR score | up to 5 minutes from delivery
  Comparison of the 1 minute and 5 minute APGAR score that the neonates received, between the groups.
The rate of prolonged second stage | immediately after completion of the delivery.
  The percentage of patients, in each group, that were defined with a prolonged second stage. The definition is more than 2 hours from complete cervical dilation until delivery of the baby in multipara patients and more than 3 hours from complete cervical dilation until delivery of the baby in nullipara patients.

CONTACTS AND LOCATIONS:
Overall Officials: Hanoch Schreiber, MD, Principal Investigator — Clalit Health Services
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: Yes
All primary and secondary outcome measures will be made available within 6 months of syudy completion